CLINICAL TRIAL: NCT06953934
Title: Mass Balance Study of [14C] ABBV-932 Following Single Oral Dose Administration in Healthy Male Volunteers
Brief Title: A Mass Balance Study of Oral [14C] ABBV-932 in Healthy Adult Male Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M24-991
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-932

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-932 (Experimental): Participants will receive a single oral dose of ABBV-932 on day 1.
  Interventions: Drug: ABBV-932

INTERVENTIONS:
Drug: ABBV-932 — Oral Capsule

SUMMARY:
The main objective of this study is to assess the safety and tolerability of ABBV-932 in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 to ≤ 29.9.0 kg/m^2 after rounding to the tenths decimal. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Male participant who is not considering fathering a child or donating sperm during the study and for 100 days after the study drug administration
* A condition of general good health, based upon the results of a medical history, physical exam

Exclusion Criteria:

* Has not participated in another [14C] absorption, distribution, metabolism, excretion (ADME) study with a radiodose above 0.1 MBq in the period of 12 months prior to screening.
* Use of any medications/products known to alter drug absorption, metabolism, or excretion processes, within 30 days or within a period defined by 5 half-lives, whichever is longer, prior to study drug administration.
* Prior exposure to ABBV-932 or cariprazine within the past 90 days.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-10-14 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ABBV-932 | Up to approximately 86 days
  Cmax of ABBV-932
Time to Cmax (Tmax) of ABBV-932 | Up to approximately 86 days
  Tmax of ABBV-932
Terminal phase elimination rate constant (λz) of ABBV-932 | Up to approximately 86 days
  Terminal phase elimination rate constant (λz) of ABBV-932
Terminal Phase Elimination Half-Life (t1/2) of ABBV-932 | Up to approximately 86 days
  Terminal phase elimination half-life of ABBV-932
Area Under the Concentration-Time Curve From Time 0 to Time t (AUCt) of ABBV-932 | Up to approximately 86 days
  AUCt of ABBV-932
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of ABBV-932 | Up to approximately 86 days
  AUCinf of ABBV-932
Number of Participants Experiencing Adverse Events | Up to approximately 103 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-991